CLINICAL TRIAL: NCT02128971
Title: A Study to Compare the Gastrointestinal Tolerability of Ferrochel®, Sumalate®,Ferrous Fumarate, Ferrous Sulfate, Ferric Glycinate, and Placebo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albion (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM-FEB-INDO-2013-01
Record Dates: First submitted 2014-04-21; First posted 2014-05-01 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Anemia
Keywords: Iron supplement study
MeSH Terms: conditions — Anemia | interventions — bis-glycino iron II; ferrous bisglycinate; ferrous fumarate; ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Ferrochel® 90 mg (Active Comparator): Ferrochel® capsule 90 mg OD for 30 days
  Interventions: Dietary Supplement: Ferrochel® 90 mg
- Sumalate® 90 mg (Active Comparator): Sumalate® capsule 90 mg OD for 30 days
  Interventions: Dietary Supplement: Sumalate® 90 mg
- Ferrous Fumarate 90 mg (Active Comparator): Ferrous Fumarate capsule 90 mg OD for 30 days
  Interventions: Dietary Supplement: Ferrous fumarate 90 mg
- Ferrous Sulfate 90 mg (Active Comparator): Ferrous Sulfate capsule 90 mg OD for 30 days
  Interventions: Dietary Supplement: Ferrous Sulfate 90 mg
- Ferric glycinate 90 mg (Active Comparator): Ferric glycinate capsule 90 mg OD for 30 days
  Interventions: Dietary Supplement: Ferric Glycinate 90 mg
- Placebo (Active Comparator): Placebo capsule OD for 30 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ferrochel® 90 mg — Ferrochel® capsule 90 mg, administered orally once daily in the morning after breakfast, for 30 days
  Other Names: Ferrous Bisglycinate
  Arms: Ferrochel® 90 mg
Dietary Supplement: Sumalate® 90 mg — Sumalate® capsule 90 mg, administered orally once daily in the morning after breakfast, for 30 days
  Other Names: Ferrous aspartoglycinate
  Arms: Sumalate® 90 mg
Dietary Supplement: Ferrous fumarate 90 mg — Ferrous fumarate capsule 90 mg, administered orally once daily in the morning after breakfast, for 30 days
  Arms: Ferrous Fumarate 90 mg
Dietary Supplement: Ferrous Sulfate 90 mg — Ferrous Sulfate capsule 90 mg, administered orally once daily in the morning after breakfast, for 30 days
  Arms: Ferrous Sulfate 90 mg
Dietary Supplement: Ferric Glycinate 90 mg — Ferric Glycinate capsule 90 mg, administered orally once daily in the morning after breakfast, for 30 days
  Arms: Ferric glycinate 90 mg
Dietary Supplement: Placebo — Placebo capsule, administered orally once daily in the morning after breakfast, for 30 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the gastrointestinal (GI) tolerability of 5 different iron supplements (Ferrochel®, Sumalate®,ferrous fumarate, ferrous sulfate and ferric glycinate) at the same dose (90mg) and placebo.

DETAILED DESCRIPTION:
Anemia, the most common disorder of blood, is characterized by a decrease in number of red blood cells (RBCs) or less than normal quantity of hemoglobin in blood.Hemoglobin is an oxygen-carrying protein inside RBCs that transports oxygen from the respiratory organs to the rest of body. Several vitamins, minerals and nutrients are required for the development and production of RBCs, such as vitamin B12, folic acid and iron. Iron is an essential component of hemoglobin. Iron deficiency accounts for half of the anemia cases worldwide, and iron deficiency anemia is the most common nutritional disorder in the world.Iron deficiency can be the result of inadequate intake in the diet, poor absorption, the extra needs during growth or pregnancy, and blood loss. Thus, children and women are at highest risk.

Full blood count and hemoglobin measurements are used to diagnose anemia, and measurement of serum ferritin level (cutoff of 12-15 mg/l) is considered as the best single and non-invasive test for the diagnosis of iron-deficiency. Treatment of anemia depends on the cause and the severity. Oral iron supplement is the simplest and most cost-effective option to treat anemia and replenish body storage.

The objective of this clinical trial is to compare the gastrointestinal (GI) tolerability of 5 different iron supplements (Ferrochel®, Sumalate®,ferrous fumarate, ferrous sulfate and ferric glycinate) at the same dose (90mg)and placebo. The primary objective is to compare the gastrointestinal tolerability of the above quoted products through:

* Self-assessment questionnaires - Gastrointestinal Symptoms Questionnaire5
* Self reported diaries

The Secondary objective of the study is to assess the change from baseline of the parameters below:

* Hemoglobin level
* Hematocrit level
* Ferritin level

This prospective clinical trial is a single-center, six-arms, randomized, double-blinded, parallel study. Subject will be screened according to inclusion exclusion criteria, and blood sample will be collected to ensure the hemoglobin and ferritin levels. Subject also will be asked to complete the Gastrointestinal Symptoms Questionnaire. The study product will be administered 30 days, orally once daily in the morning after breakfast. The study plan as follow:

Visit 1: Screening / Baseline (day -7)

1. Protocol information will be given by the investigator to potential subjects. Each participant will sign a consent form that further explains what is entailed by participating in the study as well as providing subjects with information on how to report any adverse events (AEs) that may arise.
2. Collection of demographic information and medical history.
3. A 10-mL blood sample will be collected by venipuncture for lab analysis of hemoglobin and ferritin.
4. Subjects will complete the Gastrointestinal Symptoms Questionnaire for baseline record.
5. Subjects that meet the inclusion and exclusion criteria will be scheduled for visit 2

Visit 2: Day 0

1. PI or designee will assign an unique subject ID number to each eligible subject in ascending order; the subject ID corresponds to an assigned investigational product code on the subject list and to the label on the investigational product (IP) given to the subject.
2. Subjects will complete the Gastrointestinal Symptoms Questionnaire.
3. A 10-ml blood sample will be collected by venipuncture for lab analysis of hemoglobin, ferritin and hematocrit.
4. Subject diary will be dispensed.
5. The PI or designee will dispense the investigational product capsules to subjects, according to the subject list provided. Each subject will receive sufficient investigational product capsules to last for 30 days.
6. Subjects will begin to consume the investigational product capsule once a day, at the same time after breakfast, for 30 days starting on Day 1.

Visit 3: Day 15 Window period ± 2 days will be allowed for this visit

1. A 10-ml blood sample will be collected by venipuncture for lab analysis of hemoglobin, ferritin and hematocrit.
2. Subjects will bring their unused IP to the study site. Compliance will be monitored by counting the remaining investigational product capsules. The remaining IP capsules will then be returned to the subject.
3. Subjects will complete the Gastrointestinal Symptoms Questionnaire.
4. Subject's diary will be collected and new diary will be dispensed.

Visit 4: Day 30 Window period ± 2 days will be allowed for this visit

1. A 10-mlblood sample will be collected by venipuncture for lab analysis of hemoglobin, ferritin and hematocrit.
2. The PI or designee will collect any remaining investigational product. Compliance will be monitored by counting the remaining investigational product capsules.
3. Subjects will complete the Gastrointestinal Symptoms Questionnaire.
4. Subject's diary will be collected.
5. New Subject diary will be dispensed.

Visit 5: Day 37 Window period ± 2 days will be allowed for this visit

1. Subjects will complete the Gastrointestinal Symptoms Questionnaire.
2. Subject diaries will be collected.

Adverse Event and Serious Adverse Event will be recorded since the subjects begin consuming the investigational product and throughout the study. SAE should be recorded in the SAE form and reported to Sponsor or CRA within 24 hours. All SAE will be reported to Ethic Committee and Regulatory Authority.

ELIGIBILITY:
Inclusion Criteria:

1. Women, 18-50 years of age, inclusive
2. Hemoglobin 8 g/dl - 11 g/dl
3. Ferritin levels < 20 mcg/l (20 ng/mL)
4. Subject, or subject's acceptable representative, has voluntarily signed and dated an informed consent form, approved by a local Ethics Committee/Institutional Review Board prior to any participation in the study

Exclusion Criteria:

1. Pregnant or lactating
2. Amenorrhea
3. Severe anemia (hemoglobin 7 g/dl) or other blood abnormality (e.g., leukopenia, thrombocytopenia, polycythemia vera)
4. Serious illness that may confound study results or interfere with compliance
5. Subjects that have followed specific diet, eg. high protein diet, within 30 days prior to study start
6. Subjects that have taken iron supplements within 30 days prior to study start
7. Subjects that are allergic to any of the ingredients in the products
8. Participation in other clinical trials within three months prior to screening
9. Known intolerance to oral iron supplements
10. Habitual smokers (more than 3 cigarettes per week)
11. Other medical conditions that, in the investigator's opinion, may confound study results or prelude the subject's ability to safely complete the trial

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal questionnaire to measure the gastrointestinal tolerability | change from baseline in Gastrointestinal questionnaire on 7 days after the last dose of 30 days investigational product consumption
  The gastrointestinal tolerability of the products will be assessed by self-assessment questionnaires and self-reported diaries at baseline (screening), day 0, day 15, day 30 of investigational product consumption, and 7 days after finished the investigational product.

SECONDARY OUTCOMES:
the laboratory result to measure the change from baseline | up to 30 days of investigational product consumption
  hemoglobin levels of each subject will be measured at baseline (screening), day 0, day 15 and day 30 of investigational product consumption
the laboratory result to measure the change from baseline | up to 30 days of investigational product consumption
  Hematocrit levels of each subject will be measured at baseline (screening), day 0, day 15 and day 30 of investigational product consumption
the laboratory result to measure the change from baseline | up to 30 days of investigational product consumption
  Ferritin levels of each subject will be measured at baseline (screening), day 0, day 15 and day 30 of investigational product consumption

CONTACTS AND LOCATIONS:
Overall Officials: Yahdiana Harahap, Professor, Principal Investigator — Laboratory Faculty of Pharmacy, Universitas Indonesia
Locations (1):
- Laboratory Faculty of Pharmacy, Universitas Indonesia, Depok, West Java, Indonesia